CLINICAL TRIAL: NCT04479722
Title: Safety And EFficacy of Using LEft Atrium APpendage Closure in Nonvalvular AtRial FibrillatiOn PatienTs With High Risk of ischEmiC sTroke -- A Prospective Multicenter Randomized Clinical Trial
Brief Title: Using Left Atrium Appendage Closure in NVAF Patients With High Risk of Ischemic Stroke
Acronym: SAFE-PROTECT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort Medical (Group) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SAFE-PROTECT
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-09

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: LAAC; NVAF; ischemic stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Ischemic Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microport CardioAdvance LAAC system (Experimental): Subject implant Microport CardioAdvance LAAC system to occlude LAA through percutaneous intervention.
  Interventions: Device: Left atrial appendage closure procedure
- Watchman LAAC system (Active Comparator): Subject implant Watchman LAAC system to occlude LAA through percutaneous intervention.
  Interventions: Device: Left atrial appendage closure procedure

INTERVENTIONS:
Device: Left atrial appendage closure procedure — Implant LAAC system in LAA through percutaneous intervention

SUMMARY:
To evaluate the safety and efficacy of using Microport CardioAdvance Left Atrium Appendage Closure for preventing stroke in Non-valvular atrial fibrillation (NVAF) patients who have contraindications for long-term anti-coagulation. And to support registration approval from National Medical Products Administration (NMPA).

DETAILED DESCRIPTION:
SAFE-PROTECT trial is composed of Roll-in group, small-size group and RCT group. This trial is planned to conduct in about 20 sites from China.

Roll-in group plans to enroll at most 3 subjects each site to implant experimental device for exploration and observation.

RCT group plans to enroll no less than 210 subjects who meet the inclusion/exclusion criteria, and 1:1 randomly allocated to experimental arm or comparator arm.

ELIGIBILITY:
Inclusion Criteria:

* Non valvular atrial fibrillation subjects aged ≥18 and ≤80;
* High risk of ischemic stroke: CHA2DS2VASc score ≥ 2 ( ≥ 3 for female) together with any of the following circumstances:

  1. With a recorded history (happened earlier than 6 months from now) of bleeding (including gingival/nasal/oral bleeding, skin &soft tissue bleeding, gastrointestinal bleeding, urinary tract bleeding, cerebral haemorrhage, etc.) or bleeding tendency;
  2. Intolerance or rejection of long-term anti-coagulation therapy;
  3. Suffering stroke or embolism despite routine anti-coagulation therapy;
  4. With a predicting HAS-BLED score ≥3.
* Subjects (or his/her legal representatives) are able to understand the study objectives, willing to cooperate with procedure and follow-up. Subjects who voluntarily participate in this trial and have signed the written informed consent form.

Exclusion Criteria:

* Subjects with atrial fibrillation (AF) caused by rheumatic valvular disease, moderate to severe mitral stenosis, severe mitral regurgitation, severe aortic valve disease or severe left ventricular outflow tract obstruction with pressure difference greater than 40mmHg;
* Suffering with other disease(s) requiring long-term oral anticoagulation treatment;
* Initial untreated AF, or secondary AF with clear cause (such as hyperthyroid heart disease);
* Intracardiac thrombus (including left and/or right atrium) found or persisted;
* Suffered with myocardial infarction within 3 months;
* History of previous atrial septum repair operation or Atrial Septal Occluder implantation;
* History of previous heart valve (mechanical valve) replacement operation;
* Subjects undergoing heart transplant operation;
* Subjects with symptomatic carotid artery disease (such as carotid stenosis > 50%) or subjects with vulnerable carotid artery plaque.
* Suffered with ischemic stroke or TIA recently (within 30 days);
* Known complex active atherosclerotic plaque(s) in the descending aorta or aortic arch;
* Severe heart failure (NYHA Grade Ⅳ);
* The investigator assessed that there were abnormal result(s) with clinical significance in the routine blood test of subjects；
* Severe renal abnormal: serum creatinine >250μmol/l; or on dialysis;
* Allergic or contraindicated to aspirin, clopidogrel, heparin, contrast agent, and nitinol alloy;
* Subjects who are scheduled to receive operation within 1 year after procedure, and need to stop anti-thrombotic therapy;
* Pregnant or breast-feeding subjects, or subjects who plan to have a child within 1 year after procedure;
* Subjects with a life expectancy less than 12 months;
* Subjects who are participating in another investigational drug or device clinical trial in which the primary endpoint is still not reached before enrolment;
* Subjects have other reasons that cannot maintain 2 months anticoagulation or 6 months dual antiplatelet therapy;
* Subjects with poor compliance (judged by investigator) or cannot complete the study according to the protocol due to other reasons;
* Subjects who are unsuitable to receive LAA occlusion treatment (judged by investigator).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 210 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical success | 12-month
  Freedom from ischemic stroke, hemorrhagic stroke, systemic embolism, cardiovascular death and unexplained death

SECONDARY OUTCOMES:
LAA occlusion success | 12-month
  TEE examination showing that the residual shunt < 5mm jet width or complete occlusion of LAA

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zheng, Prof., Study Chair — MicroPort Orthopedics Inc.
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices) will be shared. Additionally, study protocol will be available. The data will become available for the beginning 3 months and ending 5 years following article publication.
  If the data sharing plan changes after registration, this should be reflected in the statement submitted and published with the manuscript, and updated in the registry record.
Supporting Information: Study Protocol
Time Frame: For the beginning 3 months and ending 5 years following article publication
Access Criteria: (with) Researchers who provide a methodologically sound proposal. (For the analysis) To achieve aims in the approved proposal. (Requisite mechanism) Proposals should be directed to mzheng@microport.com. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link to be included).